CLINICAL TRIAL: NCT01801163
Title: A Phase Ib Study of Stereotactic Radiotherapy (SBRT) Plus Sorafenib in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: A Phase Ib Study of Stereotactic Body Radiotherapy (SBRT) Plus Sorafenib in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial had no patients accrued while open
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IUCRO-0404; IRB #1211009970
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Radiosurgery

ARMS (1):
- Sorafenib plus Stereotactic Radiotherapy (Experimental): Single agent Sorafenib x 2 weeks followed by Stereotactic Radiotherapy, then Sorafenib until disease progression.
  Interventions: Drug: Sorafenib; Radiation: Stereotactic radiotherapy

INTERVENTIONS:
Drug: Sorafenib — Sorafenib x 2 weeks followed by Stereotactic Radiotherapy and then sorafenib until disease progression.
Radiation: Stereotactic radiotherapy — Sorafenib x 2 weeks followed by Stereotactic Radiotherapy then Sorafenib until disease progression.

SUMMARY:
This is a research study of a radiation treatment called stereotactic body radiotherapy (SBRT) plus a medicine called sorafenib. The purpose of this study is to evaluate the safety of SBRT plus Sorafenib to see what effects (good and bad) it has on the treatment of liver cancer.

ELIGIBILITY:
Inclusion Criteria:

4.1.1Age ≥ 18 years. 4.1.2 Patients with HCC without cirrhosis or with CTP class A (maximum score 6).

4.1.3 Patient must not be a surgical candidate at presentation. 4.1.4 Able to undergo contrast enhanced MRI of the primary tumor using the liver MRI protocol.

4.1.5 Measurable disease per mRECIST criteria defined as lesions >/=1cm showing intratumoral arterial enhancement in contrast-enhanced CT or MRI and being suitable for repeat measurements.

4.1.6 Must not have evidence of metastatic disease. 4.1.7 Karnofsky performance status >/=70% 4.1.8 Life expectancy ≥ 3 months as determined by the treating physician. 4.1.9 If single tumor, maximum tumor diameter must be </= 6 cm. 4.1.10 No more than three discrete liver lesions, with the overall sum of diameters being </= 6 cm.

4.1.11 None of the lesions to be treated can be in closer than 0.5 cm to the wall of the stomach, duodenum, or hepatic flexure of the colon.

4.1.12 Radiotherapy treatment planning confirms one of the following:

* One third of the uninvolved liver should receive </=10 Gy
* At least 500 cc of uninvolved liver should receive </=7 Gy 4.1.13 Radiotherapy treatment planning confirms all of the following parameters for other normal tissues tolerance:
* Maximal cord dose: 600 cGy per fraction x3 for a total of 18 Gy.
* Right kidney: <2/3 of the kidney volume receives > 15 Gy total dose and
* Left Kidney: < 1/3 receives > 15 Gy total dose. 4.1.14 Must fit in the stereotactic body immobilization device as per institutional or manufacturer guidelines.

4.1.15 Patients must have adequate liver function within 2 weeks of study registration. Adequate liver function is defined as all of the following:

* total bilirubin < 3mg/dL
* albumin >/= 2.5 g/dL
* INR </= 1.5 and
* no greater than mild elevation of transaminases (AST, ALT < 5 x ULN) 4.1.16 Patients must have adequate renal function within 2 weeks of study registration. Adequate renal function is defined as one of the following:
* creatinine < 1.8 mg/dl or
* creatinine clearance (CrCL) >/= 50 ml/min. 4.1.17 Adequate bone marrow reserve within 2 weeks of study registration, defined as all of the following:
* ANC count >/=1500 mm3
* Platelets >/=50,000/mm3
* Hemoglobin > 9g/dL 4.1.18 No history of atherosclerotic coronary artery disease that required bypass surgery, unless 1) bypass surgery occurred more than 12 months prior to enrollment, and 2) disease is stable (in consultation with a cardiologist).

4.1.19 Women must not be pregnant or breastfeeding. The effects of Sorafenib on the developing human fetus are unknown. For this reason and because radiation therapy and Sorafenib used in this trial are may be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

4.1.20 No history of HIV positivity, as the effects of sorafenib combined with radiation therapy on patients with HIV are unknown. Patients with known HIV risk factors (as determined by the treating physician) will be not eligible for this study without HIV testing.

4.1.21 Must be able to provide written informed consent and HIPAA authorization.

Exclusion Criteria:

4.2.1 Medical history of systemic lupus erythematous, rheumatoid arthritis, systemic sclerosis or scleroderma.

4.2.2 Prior radiation therapy to the abdomen 4.2.3 Prior treatment with Sorafenib or other Ras or VEGF pathway inhibitor. 4.2.4 Minor surgical procedure (e.g fine needle aspiration or needle biopsy) within 7 days of study registration.

4.2.5 Major surgical procedure, significant traumatic injury, or serious non-healing wound, ulcer or bone fracture within 21 days of study registration; investigator has to document adequate healing has occurred prior to study registration.

4.2.6 Any of the following within 6 months prior to study drug administration: severe/unstable angina (angina symptoms at rest), new onset angina (began within the last 3 months) or myocardial infarction, congestive heart failure, cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.

4.2.7 History of thrombotic or embolic events such as cerebrovascular accident or transient ischemic attack within the past 6 months.

4.2.8 History of aneurysm or arteriovenous malformation. 4.2.9 Active, clinically serious infection >/= CTCAE grade 2. 4.2.10 Receipt of any investigational agent within 4 weeks of study registration.

4.2.11 Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management 4.2.12 Pulmonary hemorrhage/bleeding event ≥CTCAE Grade 2 within 4 weeks of study registration 4.2.13 Any other hemorrhage/bleeding event including esophageal variceal bleeding >/= CTCAE Grade 3 within 4 weeks of study registration.

4.2.14 Evidence or history of bleeding diathesis or coagulopathy 4.2.15 Chronic, daily treatment with nonsteroidal anti-inflammatory medications. (Daily aspirin use is permitted) 4.2.16 Use of carbamazepine (Carbatrol, Epitol, Equetro, Tegretol), rifabutin (Mycobutin), rifampin/ rifampicin (Rifadin, Rimactane), or ritonavir (Norvir).

4.2.17 Known or suspected allergy to Sorafenib or any agent given in the course of this trial.

4.2.18 Any condition that impairs patient's ability to swallow whole pills. 4.2.19 Any malabsorption problem that would impair the patient's ability to absorb oral medication.

4.2.20 Other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-02; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Start of sorafenib through disease progression, an expected average of 12 months.
  Adverse events will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

SECONDARY OUTCOMES:
Number of patients with local response | Start of sorafenib through disease progression, an expected average of 12 months
  The local response rate, local clinical benefit rate,and local tumor shrinkage rate (LCR+LPR+LSD's)will be tabulated. Response will be measured according to a modification of the Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Time from the start of the treatment until the criteria for overall disease progression is met or death occurs. | Start of sorafenib through disease progression, an expected average of 12 months.
Time from start of treatment until death from any cause or date of last patient contact. | Start of soafenib until death.

OTHER OUTCOMES:
3.2.3 Evaluate pharmacodynamic changes in tumor vascular parameters (e.g blood flow, blood volume, and time to peak in ROC (receiver operator characteristics curve) by DCE-MRI and correlate with efficacy outcomes | Baseline to disease progression
3.2.4 To evaluate biologic markers such as VEGF, eNOS and HIF1-alpha, VEGF-R2 genetic polymorphisms as well as serum VEGF and soluble VEGFR2 levels and correlate with efficacy outcomes. | Baseline to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Higinia Cardenes, MD PHD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States